CLINICAL TRIAL: NCT02746016
Title: Effect of Formula Supplemented With Oligosaccharides on Infant Behavior
Brief Title: Effect of Formula on Infant Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AL19
Record Dates: First submitted 2016-04-13; First posted 2016-04-21 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Gastrointestinal Tolerance
MeSH Terms: interventions — Oligosaccharides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infant Formula supplemented with Oligosaccharides (Experimental): Ready to feed infant formula ; Feed ad libitum.
  Interventions: Other: Infant Formula supplemented with Oligosaccharides

INTERVENTIONS:
Other: Infant Formula supplemented with Oligosaccharides — sole source nutrition

SUMMARY:
This is a prospective, multi-center, single-arm study to evaluate the symptoms of formula intolerance in healthy term infants.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health as determined from subject's medical history by parent report
* Subject is a singleton full-term birth with a gestational age of 37 - 42 weeks
* Subject's birth weight was ≥ 2490 g (~5 lbs. 8 oz.)
* Subject is between 7 and 42 days of age
* Infant was identified by parents as very fussy or extremely fussy in the baseline tolerance evaluation
* Infant is exclusively formula-fed at time of study entry
* Parent(s) confirm their intention not to administer vitamin or mineral supplements, solid foods or juices to their infant from enrollment through the duration of the study
* Subject's parent(s) has voluntarily signed and dated an informed consent form (ICF) prior to any participation in the study

Exclusion Criteria:

* An adverse maternal, fetal or subject medical history that has potential for effects on tolerance, growth, and/or development
* Subject is taking and plans to continue medications, home remedies, herbal preparations or rehydration fluids that might affect gastrointestinal (GI) tolerance
* Subject participates in another study that has not been approved as a concomitant study
* Subject has been fed any formula containing human milk oligosaccharides prior to study enrollment
* Subject has been treated with oral antibiotics within 7 days prior to study enrollment
* Mother intends to use a combination of breast and formula feeding

Ages: 7 Days to 42 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Fussiness | Change from baseline (3 days prior to SD1) to within one day of initiation of study feeding (SD1)
  Parent Questionnaires

SECONDARY OUTCOMES:
Fussiness | Baseline to SDAY 29
  Parent Questionnaires
Hours of daily crying | Baseline to SDAY 29
  Parent Questionnaires
Gastrointestinal Tolerance | Baseline to SDAY 29
  Parent Questionnaires
Stool Pattern | Baseline to SDAY 29
  Parent Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Borschel, PhD, RD, Study Chair — Abbott Nutrition
Locations (13):
- United States (13):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Watching Over Mothers and Babies, Tucson, Arizona
  - Norwich Pediatric Group, PC, Norwich, Connecticut
  - Florida Institute for Clinical Research, LLC, Orlando, Florida
  - Score Physician Alliance, LLC, St. Petersburg, Florida
  - Women's Clinic of Lincoln, PC, Lincoln, Nebraska
  - Institute of Clinical Research, LLC, Cleveland, Ohio
  - Aventiv Research, Grove City, Ohio
  - Coastal Pediatric Research, Charleston, South Carolina
  - DCOL Center for Clinical Research, Longview, Texas
  - Southwest Children's Research Associates, P.A., San Antonio, Texas
  - Tanner Clinic, Layton, Utah

IPD SHARING:
Plan to Share IPD: Undecided